CLINICAL TRIAL: NCT06236191
Title: Improving Sleep of Children With Neurodevelopmental Disorders: A Prospective, Randomised Controlled Trial Using Pulsed Current Stimulation Versus Melatonin
Brief Title: Improving Sleep of Children With Neurodevelopmental Disorders: Pulsed Current Stimulation Versus Melatonin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Ng Zhi Min, Principal Investigator, KK Women's and Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/2216
Record Dates: First submitted 2023-07-31; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Insomnia; Neurodevelopmental Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neurodevelopmental Disorders | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Crossover trial using Balaam's design
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor assessing sleep data will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention group is transcranial pulse electrical stimulation
  Interventions: Device: transcranial pulsed current stimulation
- Comparator (Active Comparator): comparator is Melatonin
  Interventions: Drug: Melatonin

INTERVENTIONS:
Device: transcranial pulsed current stimulation — A form of transcranial electrical stimulation that delivers unidirectional monophasic rectangular pulses of current.
  Arms: Intervention
Drug: Melatonin — Melatonin
  Arms: Comparator

SUMMARY:
This is a prospective, randomised controlled trial that evaluates whether transcranial pulsed current stimulation increased total sleep time in children with neuroevelopmental disorder, compared to Melatonin

DETAILED DESCRIPTION:
Background: Children with neurodevelopmental disorder such as cerebral palsy (CP) and autistic spectrum disorder have poor sleep. Poor sleep in these children may lead to worsening spasticity, increased caregiver burden and poorer quality of life. Use of Melatonin is a common treatment for sleep but it is not helpful in sleep maintenance. More sedating pharmacological options have side-effects if given long-term. A safe and non-invasive intervention that can improve sleep in children with neurodevelopmental disorder is needed. In recent years, non-invasive brain stimulation such as transcranial electrical stimulation (TES) has emerged as a potential treatment to improve sleep in adult patients with major depressive disorders, bipolar disorders, migraine and Parkinson's disease. Transcranial pulsed current stimulation (tPCS) is a form of TES that has increasingly gained attention as a novel safe and cost-effective treatment modality for spasticity in children with CP and for improvement of gait in adults with Parkinson's Disease.

Hypothesis: tPCS is effective in improving total sleep time (TST) in children with neurodevelopmental disorder.

Aim: We aim to objectively evaluate whether tPCS can increase TST in children with neurodevelopmental disorder, compared to Melatonin.

Methodology and Analytical approach: Based on 80%power, alpha 0.05 and 20%drop-out rate, this is a single centre randomized control, crossover trial using Balaam's design that enrols 40 children with neurodevelopmental disorder: Patients will be treated with home-based tPCSor Melatonin over 8 weeks. All patients will do sleep actigraphy and sleep questionnaire using the Sleep Disturbance Scale for Children at baseline and at the end of trial.

Clinical Significance: tPCS could serve as a potential alternative for pharmacotherapy in treatment of insomnia in children with neurodevelopmental disorders. This could change clinical practice and improve quality of care for these children.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4-16
* Neurodevelopmental disorder including cerebral palsy, autistic spectrum disorder, neurogenetic syndrome.
* Patients whose pre-intervention sleep questionnaire total score more than 46 and/or pre-intervention sleep questionnaire T-score more than 70 in any sleep domain
* Children agree to tPCS as per procedure and consent to the study, including need to shave hair at the site of stimulation at the occiput
* Parents/carers agree to tPCS as per visit schedule and procedure
* Medical practitioner's approval

Exclusion Criteria:

* History of uncontrolled epileptic disorders and seizures, brain tumours or trauma and mental diseases, substance abuse or dependence, use of benzodiazepines, neuroleptic, serotonin or dopaminergic drugs, presence of metal/ electronic implant in brain/ body eg. shunt, cochlear implant, pacemaker or defibrillator, untreated known obstructive sleep apnoea or another previously diagnosed sleep disorder, and current involvement in other tDCS or rTMS trials. Patients with history of drug allergy to Melatonin will also be excluded.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Total sleep time (TST) | 4 weeks
  Improvement in TST; the higher the TST the better

SECONDARY OUTCOMES:
Sleep latency (SL) | 4 weeks
  Reduction in sleep latency (min); the lower the sleep latency the better
Sleep efficiency (SE) | 4 weeks
  Increase in sleep efficiency (%); the higher the sleep efficiency the better
wake after sleep onset (WASO) | 4 weeks
  Reduction in WASO; the lower the WASO the better
Total score in sleep questionnaire | 4 weeks
  Reduction in total score in sleep questionnaire; max score 130 minimum score 26; the lower the better

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Min Ng, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KKWCH, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Sleep data including TST, SL, SE, WASO can be shared

DOCUMENTS (1):
  • Study Protocol (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT06236191/Prot_000.pdf